CLINICAL TRIAL: NCT03976674
Title: Evaluation of a Preoperative Cognitive Behavioural Therapy (CBT) Program Based on Self-determination Theory for Bariatric Surgery Candidates : an Open-label Controlled, Randomized, Superiority Study
Brief Title: A Preoperative Cognitive Behavioural Therapy Program Based on Self-determination Theory for Bariatric Surgery Candidates
Acronym: ACRoBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC-P0061
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery Candidate; Obesity
Keywords: Bariatric Surgery Candidate; Cognitive and Behavioural Emotional Therapies; Obesity
MeSH Terms: conditions — Obesity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients in preparation for bariatric surgery (Experimental): Patients in preparation for bariatric surgery in the endocrinology department will follow a cognitive behavioural therapy
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Control group (No Intervention): Standard practice

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — 5 group sessions (2h30/session) before the surgery
  Arms: Patients in preparation for bariatric surgery

SUMMARY:
The objective of this study is to evaluate the impact of a pre-surgical intervention program based on Cognitive and Behavioural Emotional Therapies, on the degree of dietary restriction of patients who are candidates for bariatric surgery in order to increase the long-term effectiveness of this kind of surgery

ELIGIBILITY:
Inclusion Criteria:

* Patient starting a preparation for bariatric surgery in the endocrinology department at St Philibert Hospital
* 18 ≤Age≤60 years
* Patient meeting the criteria of the High Authority of Health (HAS) for the agreement of a bariatric treatment
* Patient affiliated to the social security
* Patient giving informed consent

Exclusion Criteria:

* Low level of comprehension of French
* Pregnant women
* Patient under guardianship or curatorship.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination-Questionnaire (EDE-Q) score | One year after therapy
  The EDE-Q is a 28 item self-report questionnaire. It concerns behaviors over a 28-day time period and retains the scoring system of 0-6: 0 = behaviour was absent and 6 = behaviour was present daily or to an extreme degree

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia CHEROUTRE, Study Chair — GHICL
Locations (1):
- • Lille Catholic University Hospital Group, Saint Philibert Hospital, Lomme, Haits de France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheroutre C, Guerrien A, Rousseau A. Contributing of Cognitive-Behavioral Therapy in the Context of Bariatric Surgery: a Review of the Literature. Obes Surg. 2020 Aug;30(8):3154-3166. doi: 10.1007/s11695-020-04627-9. PMID 32440777